CLINICAL TRIAL: NCT00308100
Title: A Multicenter, Randomized, Open-Label, Parallel-Group, Albumin-Controlled Phase IV Study to Evaluate the Efficacy and Safety of Hydroxyethyl Starch (130/0.4) for Intravascular Volume Therapy in Patients Undergoing Liver Transplantation
Brief Title: Hydroxyethyl Starch (130/0.4) for Intravascular Volume Therapy in Liver Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is prematurely ended due to poor patient recruitment rate.
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Professor Leng Xisheng, Beijing Renmin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFP502
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Intraoperative Complications
Keywords: Liver Transplantation
MeSH Terms: conditions — Intraoperative Complications | interventions — Hydroxyethyl Starch Derivatives; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Hydroxyethylstarch 130/0.4
- 2 (Active Comparator)
  Interventions: Drug: 5% Albumin

INTERVENTIONS:
Drug: Hydroxyethylstarch 130/0.4 — HES 130/0.4, administered intra- and perioperatively, max. daily dose: 33ml/kg BW; if needed, additionally albumin is administered (ratio crystalloid to colloid= 1:1)
  Other Names: HES 130/0.4; Hydroxyethyl starch 130/0.4
  Arms: 1
Drug: 5% Albumin — 5% albumin, administered intra- and perioperatively
  Arms: 2

SUMMARY:
There are no standardized plasma volume replacement protocols during liver transplantation surgery. The current study is designed to compare efficacy, safety, and costs of perioperative volume replacement with Voluven (Hydroxyethyl starch 130/0.4) and albumin in patients undergoing liver transplantation.

DETAILED DESCRIPTION:
End-stage liver disease is one of the major diseases leading to death. With advancement of transplantation surgery and perioperative anesthesia management, liver transplantation has become an effective method to recover patients' liver function, thus saving their lives and improving their quality of life. Serious disorders of fluid balance, such as blood coagulation dysfunction, electrolyte disequilibrium, hypoalbuminaemia, low hematocrit, low hemoglobin and acid-base imbalance etc. exist in end stage cirrhosis patients with liver transplantation. Such abnormalities in the internal milieu could cause or worsen cardiovascular and pulmonary dysfunction, thus making perioperative management more difficult.

Albumin and blood plasma are conventionally used as plasma volume expanders in clinical practice. At the same time, the level of albumin concentration is also used as an important criterion of prognosis. When the level of albumin concentration in serum is below 35 g/L, postoperative mortality rates and complications will increase significantly. In fact, it has been the focus of debate for many years whether albumin should be used for volume replacement in critically ill patients. Boldt and his colleagues demonstrated that albumin has little positive influence on the prognosis of critically ill patients. However, Shwe deemed albumin beneficial to critically ill patients. Simon suggested that albumin is given mainly for treating hypovolemia instead of increasing the level of albumin concentration in serum. However, at the same time, he admitted there is no advantages of albumin in comparison to other colloid solutions and, furthermore, it is more expensive.

Voluven (130/0.4) is a medium molecular weight hydroxyethyl starch (HES) produced by Beijing Fresenius Kabi Pharmaceutical Co., Ltd. It is a novel HES preparation with optimized molecular weight and molecule distribution, has a lower degree of substitution (DS) (0.4), and a narrower molecular distribution profile (C2/C6) than other available HES specifications which make it more suitable for volume replacement therapy. Some studies have revealed that Voluven (130/0.4) has a comparable efficacy with HAES-steril (average molecular weight 200.000 dalton, degree of substitution 0.5). Because of its improved pharmacological profile, Voluven (130/0.4) is used to avoid capillary vessel leakage and improve oxygenation of tissues. In addition, Voluven (130/0.4) does not accumulate in plasma or tissues even after multiple dosing (maximal dose 50 ml/kg), and has an improved HES safety profile in terms of coagulation and kidney function.

The current study is designed to assess the efficacy, safety, and pharmaceutical economics characteristic of perioperative volume replacement with Voluven (130/0.4) in patients undergoing liver transplantation compared with patients who received volume therapy with albumin. The objective of this study is to supply appropriate regimens for patients undergoing liver transplantation, considering clinical efficacy, safety, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years, male or female
* Elective liver transplantation
* United Network for Organ Sharing (UNOS) Level 2A/B or 3
* Serum albumin ≥ 30 g/L
* Comprehend all the procedures of this study
* Willing and able to give informed consent

Exclusion Criteria:

* Uncontrolled exo-hepatic malignant carcinomas
* Uncontrollable infections (including HIV infection)
* Need support of artificial liver or kidney, ventilator-dependant, coma or unstable hemodynamically
* Patients with a history of hypersensitivity to hydroxyethyl starch or albumin
* Urinary output less than 500 ml within 24 hours after operation
* Patients with intracranial bleeding
* Patients with other colloids for treating hypovolemia
* Patients with pulmonary edema
* Pregnant women or females of childbearing potential and lactating mothers
* Patients who are participating in other drug studies or who receive other investigational drugs within 30 days prior to the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hemodynamics | From pre-operative period till discharged from hospital

SECONDARY OUTCOMES:
Child-Turcotte-Pugh (CTP) score | From pre-operative period till discharged from hospital
Model for End-Stage Liver Disease (MELD) score | From pre-operative period till discharged from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Xisheng Leng, MD, Principal Investigator — People's University of Peking University
Locations (1):
- People's Hospital of Peking University, Beijing, China